CLINICAL TRIAL: NCT02492113
Title: Effects of Different PEEP Levels on Work of Breathing in Morbidly Obese Patients Prior to and After Extubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, RRT, PhD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WOBTRIAL
Record Dates: First submitted 2015-06-12; First posted 2015-07-08 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Obesity
Keywords: Mechanical ventilation; Positive end-expiratory pressure; Work of breathing; Morbidly obese
MeSH Terms: conditions — Obesity | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with BMI > 35 (Experimental): ICU patients with a BMI > 35, on pressure support ventilation, scheduled for spontaneous breathing trial for evaluation of extubation
  After recruitment maneuver and decremental PEEP trial, the "Titrated-PEEP" is identified. Patients will have two spontaneous breathing trials (SBTs) in randomized order. Either the patient will receive SBT at PEEP = 0-5 cmH2O, with PSV=0 and FiO2 unchanged; or the patient will perform an SBT at "Titrated-PEEP", with the PSV=0 and FiO2 unchanged.
  Interventions: Procedure: Positive end-expiratory pressure (PEEP); Procedure: ZEEP

INTERVENTIONS:
Procedure: Positive end-expiratory pressure (PEEP) — "Titrated-PEEP". After recruitment maneuver and decremental PEEP trial, the "Titrated-PEEP" is identified. Patients will have two spontaneous breathing trials (SBTs). In this arm, patients will have SBT at "Titrated-PEEP", with the PSV=0 and FiO2 unchanged.
Procedure: ZEEP — After recruitment maneuver and decremental PEEP trial, the "Titrated-PEEP" is identified. Patients will have two spontaneous breathing trials (SBTs). In this arm, patients will have SBT at PEEP = 0-5 cmH2O, with the PSV=0 and FiO2 unchanged.

SUMMARY:
The main purpose of this study is to define at the bedside the "Titrated-PEEP" level for obese patients that increases the likelihood of extubation and ventilator liberation.

The investigators hypothesized that a titrated level of PEEP ("Titrated-PEEP") during SBT will keep the lung recruited, maintain oxygenation, and decrease the work of breathing resulting in successful ventilator liberation. In addition, post-extubation the investigators hypothesize that these patients will require noninvasive ventilatory support in the form of CPAP at the level of "titrated-PEEP" used during the SBT.

DETAILED DESCRIPTION:
The high WOB of morbidly obese patients is associated with respiratory muscle fatigue and failure in extubation. The investigators hypothesized that the use of a titrated PEEP level prior to and after extubation might improve successful extubation rates and avoid re-intubation.

In this study, patients will be awake and ventilated in the pressure support ventilation (PSV) mode. The investigators will apply different PEEP levels to measure WOB, transpulmonary pressure and characterize the response of the respiratory system to increasing or decreasing PEEP. The "Titrated-PEEP" will be identified as the PEEP level associated with the lowest value of respiratory system elastance and an end expiratory transpulmonary pressure of 2 cmH2O. Then the participants will have two spontaneous breathing trials; one at PEEP 0-5 cmH2O, and the other at the "Titrated-PEEP" level, with PSV=0 and FiO2 unchanged. After extubation, the participants will first receive CPAP set at "Titrated-PEEP", then spontaneous breathing. Electrical impedance tomography (EIT), respiratory system mechanics and gas exchange will be recorded during the study.

The investigators believe that the real-time determination of "Titrated-PEEP" can guide the treatment of mechanical ventilation and give us a better understanding of the physiology and pathophysiology of morbidly obese patients. As a result, this study will improve patient safety; reduce the duration of mechanical ventilation, complications and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated;
* Weaning from mechanical ventilation;
* BMI ≥ 35 kg/m2 with waist circumference > 88 cm for women; waist circumference > 102 cm for men.
* A well functioning arterial line.

Exclusion Criteria:

* Known presence of esophageal varices
* Recent esophageal trauma or surgery
* Severe thrombocytopenia (PTL ≤ 5,000/mm3)
* Severe coagulopathy (INR ≥ 4)
* Presence of pneumothorax
* Pregnancy
* Pacemaker and/or internal cardiac defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2015-11; Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Differences in WOB at titrated PEEP levels vs. ZEEP level | 24 hours
  Work Of Breathing measured as J/L and J/min during a Spontaneous Breathing Trial at titrated PEEP vs. Work Of Breathing measured as J/L and J/min during a Spontaneous Breathing Trial at zero PEEP

SECONDARY OUTCOMES:
Gas Exchange - Oxygenation | 24 hours
  Difference in oxygenation as measured in mmHg of PaO2/FiO2 during a Spontaneous Breathing Trial at titrated PEEP and at zero PEEP.
Gas Exchange - Arterial carbon dioxide | 24 hours
  Difference in arterial carbon dioxide as measured in mmHg (PaCO2) during a Spontaneous Breathing Trial at titrated PEEP and at zero PEEP.
Respiratory Mechanics - Compliance | 24 hours
  Difference in Compliance, measured as ml/cmH2O, of the respiratory system, lungs and chest wall during a Spontaneous Breathing Trial at titrated PEEP and at zero PEEP.
Gas Volume Distribution | 24 hours
  Difference in the images of Electric Impedance Tomography measured as relative variation of regional impedance (deltaZ) (i.e. distribution of ventilation) during a Spontaneous Breathing Trial at titrated PEEP and at zero PEEP.
Hemodynamics - Blood pressure | 24 hours
  Changes in arterial blood pressures (BP, mmHg) during a Spontaneous Breathing Trial at titrated PEEP and at zero PEEP.
Hemodynamics - Heart rate | 24 hours
  Changes in heart rate (HR, bpm) during a Spontaneous Breathing Trial at titrated PEEP and at zero PEEP.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kacmarek, RRT, PhD, Principal Investigator — Massachusetts General Hospital; Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachussets General Hospital, Boston, Massachusetts, United States